CLINICAL TRIAL: NCT07195058
Title: Trauma-informed Obstetric Care for Perinatal Health in Women With Histories of Childhood Abuse: a Pilot Randomized Clinical Trial
Brief Title: Trauma-informed Obstetric Care for Perinatal Health: a Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Hospital Materno Infantil Ramón Sardá (Network)
Responsible Party: Principal Investigator, Pamela Scorza, Assistant Professor of Women's Mental Health in Psychiatry, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAU8914
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Mother to Child Transmission; Breast Feeding; Trauma
Keywords: Adverse childhood experiences (ACE); Edinburgh Postnatal Depression Scale (EPDS); Perceived Stress Scale (PSS); Maternal antenatal attachment scale (MAAS); Social Support Questionnaire (SSQ); Prenatal Distress Questionnaire (NuPDQ); Iowa Infant Feeding scale (IIFAS); Trauma Informed Care
MeSH Terms: conditions — Breast Feeding; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Women will be randomized to intervention (care with clinicians trained in the TIOC model) or control (treatment as usual). Both groups will receive all study evaluations in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trauma Informed Obstetric Care (TIOC) (Experimental): Women randomized to the trauma informed obstetric care (TIOC) intervention will be scheduled for all their prenatal appointments with obstetricians trained in the TIOC model. Additionally, the midwife on duty in the delivery ward will ensure that all items on a checklist of trauma-sensitive birth practices are followed during that participant's labor and delivery
  Interventions: Behavioral: Trauma Informed Obstetric Care (TIOC)
- Treatment as usual (TAU) (No Intervention): Participants randomized to TAU will receive usual prenatal care, which includes a referral to psychological services when deemed necessary by the prenatal care provider. These participants' prenatal visits will not be scheduled with providers who have received TIOC training.

INTERVENTIONS:
Behavioral: Trauma Informed Obstetric Care (TIOC) — TIOC providers will receive a training that was developed for this study. Elements of trauma-informed care described in the literature -combined with the experience of the study team, with deep expertise in trauma-informed obstetric care, were used to create three training modules, each of which includes didactics and role-plays to help participants practice and embody skills they learn. The three modules are:
  1. Effects of trauma on physiological and psychological process relevant to pregnancy and childbirth.
  2. Body language and verbal language for safety, respect, and patient agency
  3. Recognizing and responding to distress and dissociation
  Arms: Trauma Informed Obstetric Care (TIOC)

SUMMARY:
The study will test trauma-informed obstetric care training and supervision for obstetric clinicians in relation to prenatal mental health and attachment formation (early predictors of child development) in women presenting for prenatal care in a public hospital in Buenos Aires, Argentina.

DETAILED DESCRIPTION:
Infants of women who have experienced trauma have up to five times the risk of health and developmental problems. Low-income women are more likely to experience trauma, a factor in the intergenerational transmission of racial and socioeconomic inequities in health and development. In women with trauma histories, pregnancy and the period after the baby is born can be particularly stressful. A new way of improving pregnancy and early childhood outcomes in women with trauma histories is to train obstetric clinicians in the delivery of obstetric care attuned to the unique needs of women with histories of childhood abuse. Models of trauma-informed obstetric and gynecological care (TIOC) have been developed, however, none of these TIOC models have been formally tested for effectiveness. This study aims to develop and test a model of TIOC in a public hospital in Argentina that serves women who experience a high degree of disadvantage.

ELIGIBILITY:
Inclusion Criteria:

* Women who are <19 weeks pregnant
* Nulliparous (no previous live births)
* 18 or more years of age
* Carrying a single fetus
* Can speak Spanish

Exclusion Criteria:

* Any current psychiatric diagnosis or treatment
* Medical complications (hypertension, cardiac disease, diabetes, chronic disease, autoimmune disease) before pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) Score | 8-22 weeks gestation, 28-35 weeks gestation
  Depression and anxiety symptoms during pregnancy will be measured by the EPDS. The scores range from a minimum of 0 to a maximum of 30. The total score reflects the level of depression, with higher scores indicating higher depression.
Perceived Stress Scale (PSS) Score | 8-22 weeks gestation, 28- 35 weeks gestation
  Perceived stress during pregnancy will be measured by the PSS. Scores range from a minimum of 0 to a maximum 40. The total score reflects the level of stress during pregnancy, with higher scores indicating higher stress.
Maternal Antenatal Attachment Scale (MAAS) Score | 8-22 weeks gestation, 28-35 weeks gestation
  Maternal Attachment Feelings toward fetus during pregnancy will be measured by the MAAS. Scores range from a minimum of 19 to a maximum of 95. The total score reflects maternal attachment, with higher scores indicating higher maternal-fetal attachment.
CARE Scale Score | 8-22 weeks gestation, 28-35 weeks gestation, 0-48 hours after birth
  The mother's experience of care provided will be measured by the CARE Scale. Scores range from a minimum of 10 to a maximum of 50. The total score reflects the level of perceived empathy, with higher scores indicating higher empathy.
Prenatal Distress Questionnaire (PDQ) Score | 8-22 weeks gestation, and 28-35 weeks gestation
  Pregnancy-specific distress will be measured by the PDQ. Scores range from a minimum of 0 to a maximum of 34. The total score reflects the level of prenatal distress, with higher scores indicating higher levels of prenatal stress.

SECONDARY OUTCOMES:
Childbirth Experiences Questionnaire Score | 0-48 hours after birth
  The mother's experience of childbirth will be measured with the Childbirth Experiences Questionnaire. The total score ranges from 1 to 4, with 1 indicating positive experiences of childbirth and 4 indicating negative experiences of childbirth.
Iowa Infant Feeding Attitudes Scale Score | 0-48 hours after birth
  The mother's attitudes and attention towards infant feeding will be measured using the Iowa Infant Feeding Attitudes Scale. Scores range from a minimum of 17 to a maximum 85, with a higher score indicating more positive attitudes toward breastfeeding.
Gestational Age at Birth | 0-48 hours after birth
  Infant's gestational age at birth.
Birthweight | 0-48 hours after birth
  Infant's weight at birth.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Scorza, ScD, Principal Investigator — Columbia University
Locations (1):
- Hospital Materno Infantil Ramon Sardá, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided